CLINICAL TRIAL: NCT03625375
Title: Effects of Combined Exercises on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dysmenorrhea
Record Dates: First submitted 2018-06-04; First posted 2018-08-10 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Primary Dysmenorrhea
Keywords: exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Individuals will perform exercises 3 times a week.
  Interventions: Other: Exercise
- Control Group (No Intervention): Individuals will not perform exercises

INTERVENTIONS:
Other: Exercise — Intervention consist of aerobic, stretchig, pelvic motions, kegels and relaxation exercises
  Arms: Treatment Group

SUMMARY:
Dysmenorrhea is one of the most common gynecological problem in adolescents and young women. Symptoms of dysmenorrhea include pelvic / abdominal pain, back pain, headache, nausea, vomiting, diarrhea. These symptoms occur before menstrual bleeding or with bleeding and lasts in 12-74 hours. The objective of this study to investigate the effects of combined exercises on dysmenorrhea symptoms. Exercise protocol aerobic, stretching, kegels, pelvic motions and relaxation exercises.

DETAILED DESCRIPTION:
Women with a positive primary dysmenorrhoea symptom between 18 and 30 years of age living in the Turkish Republic of Northern Cyprus will be included in the study. According to the result of the power analysis, 14 subjet for control and 14subjet intervention group were decided.

The eligibility criteria for this study are:

* The Visual Analogue Scale value is at least 5 per day when the dysmenorrhea symptoms are the most painful,
* To have the regular menstrual cycle (24-35 days),
* To be sedentary

The exclusion criteria for this study are:

* Women with secondary dysmenorrhea,
* The women who gave birth or abortion,
* People with active sexual experience,
* Women who use intrauterine devices,
* Individuals with regular drug use,
* Serious psychological problems
* Acute musculoskeletal problems,
* People with neurological or cardiopulmonary disease

This research will consist of exercise and control groups. An exercise protocol consisting of a combination of various exercises will be applied to the exercise group and no exercises will be done for the control group. women in the exercise group will perform two menstrual cycles, three times a week in the presence of a physiotherapist.

Assessments will be made on the day that the symptoms are seen to be the most severe in order to determine the symptoms of the women in both groups. After baseline assements exercises will start at 3rd day of cycle. Assesments will repeat at second and third menstrual bleedings.

Visual Analogue Scale, Menstrual symptom questionnarie and Pittsburgh Sleep Quality Index will be use.

ELIGIBILITY:
Inclusion Criteria:

* The Visual Analogue Scale value is at least 5 per day when the dysmenorrhea symptoms are the most painful,
* To have the regular menstrual cycle (24-35 days),
* Being a sedentary (not participating in any regular exercise program).

Exclusion Criteria:

* Women with secondary dysmenorrhea,
* The women who gave birth or abortion,
* People with active sexual experience,
* Women who use intrauterine devices,
* Individuals with regular drug use,
* Serious psychological problems
* Acute musculoskeletal problems,
* People with neurological or cardiopulmonary disease.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
pain changes from baseline to 8 weeks | To asses pain level changes in this study assement make at baseline and repeat after 1 and 2 months
  to asses pain level with Visual Analogue Scale. 0 means no pain. Higher points means higher pain.

SECONDARY OUTCOMES:
menstrual symptoms changes from baseline to 8 weeks | At baseline, after 4 weeks from baseline and 8 weeks after baseline
  to asses menstrual symptoms with menstrual symptoms questionnarie. we will use total point as a data. points are vary between 0 and 110. Higher points means having worse menstrual symptpms.
sleep quality changes from baseline to 8 weeks | At baseline of the study, after 4 weeks from baseline and 8 weeks after baseline
  to asses sleep quality with pittsburgh sleep quality index. We will use total point as data. lowest grade is 0 and 21 is higher point. 0-5 means good sleep, after 10 point it means worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kırmızıgil, Study Director — Eastern Meditteranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kirmizigil B, Demiralp C. Effectiveness of functional exercises on pain and sleep quality in patients with primary dysmenorrhea: a randomized clinical trial. Arch Gynecol Obstet. 2020 Jul;302(1):153-163. doi: 10.1007/s00404-020-05579-2. Epub 2020 May 15. PMID 32415471